CLINICAL TRIAL: NCT03982654
Title: Investigating the Physiology of Labour, Labour Onset and Pregnancy Outcomes in Pregnant Women, Through Longitudinal Measurements Performed With a Wearable Sensor
Brief Title: Investigating the Physiology of Labour and Labour Onset Through Longitudinal Measurements Performed With a Wearable Sensor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bloom Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: WISH01
Record Dates: First submitted 2019-05-20; First posted 2019-06-11 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2019-06

CONDITIONS: Labour Onset

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bloomlife (Experimental)
  Interventions: Device: Bloomlife

INTERVENTIONS:
Device: Bloomlife — Women use the Bloomlife sensor to collect data throughout their pregnancy. The collected data is stored locally in the device, but it is not used to provide any feedback to the patients or to the clinical team. Therefore the use of the device doesn't have an impact on clinical decision making and patients' care.

SUMMARY:
The purpose of the study is to collect data to support the development and validation of a machine learning model for the automatic detection, prediction and monitoring of labour, through the use of a wearable sensor (Bloomlife sensor) that can be easily used at home.

Women participating in the study will be asked to regularly record data with the Bloomlife sensor, from inclusion in the study until delivery. In addition, clinical information related to their pregnancy and delivery will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant
* Gestational age between 20 weeks and 0 days and 30 weeks and 0 days
* Willingness to participate in the study

Exclusion Criteria:

* Implanted pacemaker or any other implanted electrical device
* History of allergies to silicone-based adhesives
* Any health condition resulting in higher chance of C-section (meeting one of these criteria is sufficient to be excluded): previous history of C-section, placental abnormality, being primipara and older than 40

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2018-11-26 (Actual); Study Completion 2019-03-05 (Actual)

PRIMARY OUTCOMES:
Accuracy | At delivery
  Accuracy of the machine learning model for the automatic detection of labor, measured in terms of sensitivity and specificity in detecting labour

SECONDARY OUTCOMES:
Labour probability | At delivery
  Probability of being in labour, computed using electrophysiological signals collected with the Bloomlife sensor

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried Gyselaers, MD, PhD, Principal Investigator — Ziekenhuis Oost-Limburg; Frederic Chantraine, MD, PhD, Principal Investigator — CHR de la Citadelle
Locations (2):
- Belgium (2):
  - Ziekenhuis Oost-Limburg, Genk
  - CHR de la Citadelle, Liège